CLINICAL TRIAL: NCT06504849
Title: Instant Message-delivered Personalised Lifestyle Modification Intervention for Pre-hypertension Management Among Community Dwelling Adults: a Randomised Controlled Trial
Brief Title: Instant Message-delivered Personalised Lifestyle Modification Intervention for Pre-hypertension Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pre-HTN2024
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-03

CONDITIONS: Pre-hypertension; Lifestyle Modification; Blood Pressure Management; Mobile Phone Use
MeSH Terms: conditions — Prehypertension; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will receive personalised brief LSM messages (according to their unhealthy behaviours and preferences, screened during the baseline measurement) using instant messaging applications with an active self-BP monitor for 3 months. Chat-based support will also be given to the participants as an extension of the LSM messages.
  Interventions: Behavioral: Receiving LSM messages.
- Control group (Other): The control group will receive a flyer with brief pre-HTN information, which is distributed during the recruitment phase, as well as brief pre-HTN messages via instant messaging applications.
  Interventions: Behavioral: Receiving brief pre-HTN messages.

INTERVENTIONS:
Behavioral: Receiving LSM messages. — * LSM messages via instant messaging applications
  * Chat-type support messages via instant messaging applications
  Arms: Intervention group
Behavioral: Receiving brief pre-HTN messages. — * A flyer with brief pre-HTN information which is distributed during the recruitment phase
  * Brief pre-HTN messages via instant messaging applications
  Arms: Control group

SUMMARY:
To assess the effectiveness of instant message-delivered personalised lifestyle modification (LSM) intervention for pre-hypertension (pre-HTN) management among community dwelling Chinese adults.

DETAILED DESCRIPTION:
Systolic blood pressure (BP) of 120-139 or diastolic BP 80-89mmHg were previously described as 'high normal' or 'above-optimal', but have been re-defined as pre-hypertention (HTN) in the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure(JNC-7) in order to raise awareness regarding the risks of elevated BP and to emphasise healthcare professionals' roles in managing elevated blood pressures as part of primary HTN prevention. Prevalence of pre-HTN is significant, specifically reported as 36.4% of adults in a large-scale population study conducted in mainland China. Furthermore, evidence has shown that the incidence of clinical HTN over 4 years in people with pre-HTN is twice that of people with normal BP, of which approximately 17% had accelerated progression to more advanced stages of HTN. The data highlight that a significant proportion of populations at risk of developing HTN if pre-HTN remains undetected and unmanaged, and also the importance of screening for pre-HTN to initiate management and mitigate the risks associated with HTN.

Lifestyle modification (LSM) is the primary intervention for people with pre-HTN as they play a significant role in lowering BP without the use of pharmacological treatments. Both LSM interventions and pharmacological treatments have been recommended for people with HTN in clinical and public health guidelines. Ecological momentary intervention (EMI) is defined as a health intervention delivered though the mobile device's messaging functions, particularly instant messaging.In existing randomised controlled trials (RCTs), EMI also showed efficacy on LSM, including smoking cessation, diet control, psychological well-being, and weight loss. EMI can therefore serve as an important 'platform' to deliver the LSM intervention in a personalised, real-time and in-situ format.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic BP 120-139 or diastolic BP 80-89mmHg. The BP screening procedures and requirements (i.e., office BP measurement and ABPM) will strictly follow the International Society of Hypertension's Global Hypertension Practice Guidelines;
2. Aged ≥18 years;
3. Able to read and communicate in Chinese; and
4. Able to use mobile phone instant messaging function.

Exclusion Criteria:

1. Ever diagnosis of HTN;
2. Ever diagnosis of cardiovascular diseases (CVDs);
3. Pregnant or <3-month post-partum;
4. Current diagnosis of psychiatric disease or currently taking a psychotropic drug; and
5. Currently participating in any type of BP reduction intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
24hr-systolic and diastolic BP | 6 months
  The BP will be measured by 24hr-ambulatory BP monitoring.

SECONDARY OUTCOMES:
DASH diet adherence (Self-reported quesionnaire) | 6 months
  A self-reported questionnaire will be utilized to assess adherence to the DASH diet, based on the portions consumed in the previous week as reported by the participants.
Salt-intake literacy (Chinese Health Literacy Scale for Low Salt Consumption - Hong Kong, CHLSALT-HK) | 6 months
  The 49-item CHLSalt-HK had a possible score range of 0 to 98, with a higher score indicating higher health literacy related to salt intake.
Physical activity (International Physical Activity Questionnaire - Short Form, IPAQ-SF) | 6 months
  The IPAQ-SF is designed to measure the level of physical activity among adults over a week, including vigorous and moderate activities, walking, and sitting time. Scoring is based on the type, frequency, and duration of activities, converting activity levels into Metabolic Equivalent Task (MET) minutes per week to assess overall physical activity. Vigorous activities are calculated at 8 METs per minute, moderate activities at 4 METs, and walking at 3.3 METs. The total activity score is the sum of MET minutes per week for all activities, categorizing participants into low, moderate, or high physical activity levels based on their total score.
Body Mass Index (BMI) | 6 months
  BMI is calculated by dividing an individual's weight in kilograms by their height in meters squared. Higher BMI can indicate higher body fatness.
Psychological well-being (Patient Health Questionnaire, PHQ-4) | 6 months
  A 4-item scale with score ranging from 0 to 12, higher scores indicate higher severity of mental health problems.
Quality of life (EuroQol 5-dimension 5-level questionnaire, EQ-5D-5L) | 6 months
  The EQ-5D-5L assesses five health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on five levels of severity, with scores ranging from -0.864 to 1, where higher scores indicate better quality of life. Additionally, it includes a visual analogue scale (VAS), ranging from 0 (the worst health imaginable) to 100 (the best health imaginable).
Feedback on instant message-delivered personalised lifestyle modification intervention | 6 months
  Feedback on the blood pressure management program will be collected, focusing on various aspects such as perceived usefulness and willingness to recommend the program. Each aspect will be evaluated using a 5-point Likert scale, where higher scores indicate more positive evaluations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong